CLINICAL TRIAL: NCT02029391
Title: Kinesio Taping on Short Term Changes in Subjects With Myofascial Pain Syndrome: a Randomized Controlled Trial
Brief Title: Kinesio Taping in Subjects With Myofascial Pain Syndrome: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201304048RINB
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial pain syndrome; taping; manual therapies
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myofascial pain syndrome patients (Active Comparator): Manual pressure release only
  Interventions: Other: Manual pressure release
- Myofascial pain syndrome (Experimental): One session of manual pressure release and kinesio tape
  Interventions: Other: Manual pressure release; Other: Kinesio tape

INTERVENTIONS:
Other: Manual pressure release — Therapist applied non-painful pressure with slowly increase over the myofascial trigger point until he felts a tissue resistance barrier.
Other: Kinesio tape — Kinesio tape was adhered from insertion to origin of the upper trapezius muscle
  Arms: Myofascial pain syndrome

SUMMARY:
Musculoskeletal dysfunction is considered as a major public health problem affecting about one third of the adult population. Myofascial pain syndrome (MPS) characterized by myofacial trigger points as well as fascia tenderness are thought to be the main cause of musculoskeletal dysfunction. The aim of the treatment for musculoskeletal dysfunction is to reduce pain and restore normal function. Clinically, some evidence supports the application of kinesio tape in these patients. The underlying mechanism, however, is not clear. The investigators goal was to validate proposed mechanism of kinesio tape in these patients. The primary outcome are muscle stiffness, pain intensity and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 60 years
* shoulder or neck pain corresponding with the area covered by the upper trapezius muscle
* Trigger point (taut band) in the upper trapezius muscle

Exclusion Criteria:

* diagnosis of fibromyalgia syndrome
* having undergone myofascial therapy within the past month before the study
* history of cervical spine or shoulder surgery
* previous history of a whiplash injury;
* diagnosis of cervical radiculopathy or myelopathy;
* taking medicine that might change the pain intensity or pain threshold, such as analgesics, sedatives, substance abuse (including alcohol, narcotics);
* a cognitive impairment that would prevent them from being able to understand and/or participate fully in the intervention or the measures.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Muscle stiffness | baseline, immediate after intervention and at week 1

SECONDARY OUTCOMES:
Visual analog scale (VAS) | baseline, immediate after intervention and at week 1
Pressure pain threshold | baseline, immediate after intervention and at week 1

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-Jeng Lin, PhD, Study Chair — Institute of Physical Therapy, National Taiwan University
Locations (1):
- Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan, Taiwan